CLINICAL TRIAL: NCT03249506
Title: Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus
Brief Title: Cardiovascular Outcomes in Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108355; RRA-17640 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin; empagliflozin; dapagliflozin; Dipeptidyl-Peptidase IV Inhibitors; 2,4-thiazolidinedione; Sulfonylurea Compounds; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Non-SGLT2i new Users: This is a retrospective cohort study identifying participants with type 2 diabetes mellitus (T2DM) and established cardiovascular (CV) disease using the Military Health System (MHS) over a 3-year period. Cohort 1 included participants with incident exposure of one or more non-sodium glucose co-transporter 2 inhibitor (SGLT2i) anti-hyperglycemic agent (AHA) therapy during the study period with no prior or subsequent SGLT2i exposure throughout the study period. New users are defined as participants whose first exposure to any non-metformin AHA medication occurs greater than or equal to (>=) 365 days after their start of observation in the database with no prior exposure to any medication within the same AHA medication class in the prior 365 days.
  Interventions: Drug: Dipeptidyl Peptidase-4 Inhibitor (DPP-4); Drug: Glucagon-Like Peptide-1 Agonist (GLP-1); Drug: Thiazolidinedione (TZD); Drug: Sulfonylureas; Drug: Insulin
- Cohort 2: SGLT2i new Users: Cohort 2 included participants with incident SGLT2i exposure during the study period regardless of prior or concurrent exposure to one or more additional AHA therapy. New users are defined as participants whose first exposure to SGLT2i medication occurs >= 365 days after their start of observation in the database with no prior exposure to the same AHA medication class in the prior 365 days.
  Interventions: Drug: Canagliflozin; Drug: Empagliflozin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Canagliflozin — Participants who received canagliflozin as a part of routine clinical practice and met new user criteria, will be included in SGLT2i new user group.
  Groups: Cohort 2: SGLT2i new Users
Drug: Empagliflozin — Participants who received empagliflozin as a part of routine clinical practice and met new user criteria, will be included in SGLT2i new user group.
  Groups: Cohort 2: SGLT2i new Users
Drug: Dapagliflozin — Participants who received dapagliflozin as a part of routine clinical practice and met new user criteria, will be included in SGLT2i new user group.
  Groups: Cohort 2: SGLT2i new Users
Drug: Dipeptidyl Peptidase-4 Inhibitor (DPP-4) — Participants who received a DPP-4 as a part of routine clinical practice and met new user criteria, will be included in non-SGLT2i new users group.
  Groups: Cohort 1: Non-SGLT2i new Users
Drug: Glucagon-Like Peptide-1 Agonist (GLP-1) — Participants who received a GLP-1 as a part of routine clinical practice and met new user criteria, will be included in non-SGLT2i new users group.
  Groups: Cohort 1: Non-SGLT2i new Users
Drug: Thiazolidinedione (TZD) — Participants who received a TZD as a part of routine clinical practice and met new user criteria, will be included in non-SGLT2i new users group.
  Groups: Cohort 1: Non-SGLT2i new Users
Drug: Sulfonylureas — Participants who received a sulfonylureas as a part of routine clinical practice and met new user criteria, will be included in non-SGLT2i new users group.
  Groups: Cohort 1: Non-SGLT2i new Users
Drug: Insulin — Participants who received a insulin as a part of routine clinical practice and met new user criteria, will be included in non-SGLT2i new users group.
  Groups: Cohort 1: Non-SGLT2i new Users

SUMMARY:
The purpose of this study is to identify and evaluate the event rate of the composite endpoint of all-cause mortality (ACM) or hospitalization for heart failure (HF) for participants with Type 2 Diabetes mellitus (T2DM) and established cardiovascular (CV) disease among new users of sodium-glucose co-transporter 2 inhibitor (SGLT2i) as compared with new users of non-SGLT2i anti-hyperglycemic agent (AHA).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM), defined as: greater than or equal to (>=) 1 anti-hyperglycemic agent (AHA) medication in the study period, and; >=1 diagnosis of T2DM in any available diagnosis field on or prior to index
* Established cardiovascular disease, defined as >=1 diagnosis in any diagnosis field for any of the following conditions: cerebrovascular disease; coronary artery disease (including heart failure [HF]); peripheral artery disease
* >=1-year pre-index continuous eligibility; enrollment gaps of less than or equal to (<=) 30 days will be considered continuous enrollment

Exclusion Criteria:

* Type 1 Diabetes mellitus (T1DM) diagnosis on or prior to the index date
* Secondary diabetes mellitus (DM) on or prior to the index date
* Missing sex data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with type 2 diabetes mellitus (T2DM) and established cardiovascular (CV) disease using the military health system (MHS) over a 3-year period (4/01/2013 to 3/31/2016) will be observed for the cardiovascular outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 25358 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of the Composite of All-cause Mortality (ACM) or Hospitalization for Heart Failure (HF) | approximately 3 years
  Composite of ACM and hospitalization of HF will be assessed in participants with type 2 diabetes mellitus. ACM is defined as any record of death regardless of the cause of death and is identified through a master death file within the military health system (MHS) that compiles, processes, and validates all death records from the following data sources: inpatient hospitalization discharge dispositions from military and civilian hospitals, ambulatory and outpatient encounter records with recorded death disposition, casualty death feed related to active duty service member combat related deaths, survivor self-report, and an established, recurring social security death index (SSDI) feed from the social security administration. Hospitalization for HF will be defined as any inpatient hospitalization record, inclusive of both military and civilian hospitals, with an international classification of disease-9th or 10th edition (ICD-9/10) in the primary diagnosis field.

SECONDARY OUTCOMES:
Incidence Rate of All-Cause Mortality | approximately 3 years
  ACM is defined as any record of death regardless of the cause of death and is identified through a master death file within MHS that compiles, processes, and validates all death records from the following data sources: inpatient hospitalization discharge dispositions from military and civilian hospitals, ambulatory and outpatient encounter records with recorded death disposition, casualty death feed related to active duty service member combat related deaths, survivor self-report, and an established, recurring SSDI feed from the social security administration.
Incidence Rate of Hospitalization for HF | approximately 3 years
  Hospitalization for HF will be defined as any inpatient hospitalization record, inclusive of both military and civilian hospitals, with an international classification of disease-9th or 10th edition (ICD-9/10) in the primary diagnosis field.
Incidence Rate of Major Adverse Cardiovascular Events (MACE) | approximately 3 years
  MACE will be defined as the composite endpoint of ACM, non-fatal stroke, or non-fatal myocardial infarction (MI).
Incidence Rate of Composite of MACE or Hospitalization for HF | approximately 3 years
  Participants for composite of ACM and hospitalization of HF will be assessed. MACE will be defined as the composite endpoint of ACM, non-fatal stroke, or non-fatal myocardial infarction (MI). Hospitalization for HF will be defined as any inpatient hospitalization record, inclusive of both military and civilian hospitals, with an international classification of disease-9th or 10th edition (ICD-9/10) in the primary diagnosis field.
Incidence Rate of Non-fatal stroke | approximately 3 years
  Non-fatal stroke will be defined as any inpatient hospitalization record, inclusive of both military and civilian hospitals, with an ICD-9/10 in the primary diagnosis field pertaining to either ischemic stroke or hemorrhagic stroke and the participant did not die during the index hospitalization.
Incidence Rate of Non-Fatal Myocardial Infarction | approximately 3 years
  Non-fatal MI will be defined as any inpatient hospitalization record, inclusive of both military and civilian hospitals, with an ICD-9/10 in the primary diagnosis field and the participant did not die during the index hospitalization.
Percentage of Participants With Below Knee Lower Extremity (BKLE) Amputation | approximately 3 years
  The occurrence of a below-knee lower extremity amputation will be defined by observing an associated procedure code in the outpatient or inpatient medical service claims.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Health ResearchTx, LLC, Trevose, Pennsylvania, United States